CLINICAL TRIAL: NCT05308992
Title: User Preference Study of 60 Couples Using an Experimental HydroGlyde Male Condom Compared to a Commercial Latex Male Condom
Brief Title: User Preference Study of an Experimental HydroGlyde Male Condom Compared to a Commercial Latex Male Condom
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HydroGlyde Coatings, LLC (Industry)
Collaborators: Essential Access Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HGC-002
Record Dates: First submitted 2022-03-10; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Condom Users
Keywords: Condom Use; Latex condoms; Lubrication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Couples who use condom (Other): The investigator will recruit heterosexual couples who have experience using silicone-lubricated latex condoms. All couples are required to have a backup birth control option and must be monogamous to participate in the study.
  Interventions: Device: HydroGlyde Condom

INTERVENTIONS:
Device: HydroGlyde Condom — The latex HydroGlyde condom has a hydrophilic coating which maintains its lubricity when in contact with water. Improved lubrication during intercourse may lead to improved user satisfaction and increased condom use which would help prevent the spread of Sexually Transmitted Infections and unwanted pregnancies.

SUMMARY:
Latex condoms have long been available as contraceptive devices as well as an effective means of preventing the spread of sexually transmitted infections. However, lack of adequate lubrication leads to inconsistent and incorrect condom use. The latex HydroGlyde condom has a hydrophilic coating which maintains its lubricity when in contact with water. Improved lubrication during intercourse may lead to improved user satisfaction and increased condom use which would help prevent the spread of Sexually Transmitted Infections and unwanted pregnancies.

The primary objective of this study is to evaluate the preference, performance (breakage, slippage), safety (adverse events) and acceptability of a HydroGlyde prototype condom compared to a commercial latex condom with silicone lubricant. A secondary objective of this study is to compare and evaluate various lubricant activation methods for reliability, usability, and user preference.

DETAILED DESCRIPTION:
Latex condoms have long been available as contraceptive devices as well as an effective means of preventing the spread of sexually transmitted infections. However, lack of adequate lubrication leads to inconsistent and incorrect condom use. The latex HydroGlyde condom has a hydrophilic coating which maintains its lubricity when in contact with water. Improved lubrication during intercourse may lead to improved user satisfaction and increased condom use which would help prevent the spread of Sexually Transmitted Infections and unwanted pregnancies.

The primary objective of this study is to evaluate the preference, performance (breakage, slippage), safety (adverse events) and acceptability of a HydroGlyde prototype condom compared to a commercial latex condom with silicone lubricant. A secondary objective of this study is to compare and evaluate various lubricant activation methods for reliability, usability, and user preference.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 45 years (inclusive)
2. Willing and able to give signed informed consent.
3. Willing to respond to questions concerning their reproductive and contraceptive history and use of condoms contained on self-administered questionnaires, online questionnaires or in-person interviews.
4. Have vaginal intercourse at least once weekly.
5. Protected against pregnancy by oral contraceptives, an intrauterine device, an implant, contraceptive injections, contraceptive patch, or sterilization (tubal ligation or vasectomy).
6. Willing to use the study products for four acts of vaginal intercourse within three weeks of study entry.
7. In a mutually monogamous relationship with their study partner for at least 6 months and be willing to remain mutually monogamous throughout study participation.

i. Agree not to wear any genital piercing jewelry or use sex toys while using the study condoms.

j. Agree not to use drugs that could enhance or diminish sexual response, including testosterone, poppers, and drugs like Viagra and Cialis when using study condoms.

k. Agree not to use alcohol in amounts that could enhance or diminish sexual response when using the condoms.

l. Agree to return any unopened condoms m. Have home access to the internet, a valid personal email for each partner and be reachable by mobile phone.

n. Willing to participate in either in-person visits or remote study visits conducted via videoconference and telephone and curbside exchange.

o. Agree to complete online questionnaires after testing each study product and group of study products.

p. Male partner agrees to ejaculate during vaginal intercourse. q. Willing to complete interviews by phone or video with HydroGlyde Coatings representatives.

r. Each partner has used 10 or more male condoms in their lifetime. s. Willing to sign a confidentiality agreement pertaining to the study condoms.

Exclusion Criteria:

1. Currently participating in another clinical study.
2. Female partner self-reported as pregnant.
3. Allergic to natural rubber latex or has a history of recurrent adverse events following use of latex products.
4. Known allergy or skin sensitivity to common cosmetics and/or contact lens solutions or polyvinylpyrrolidone (PVP).
5. Unable to follow instructions or strictly adhere to the study schedule.
6. At significant (high) risk of sexually transmitted infections, including human immunodeficiency virus infection, or having a medical history of recurrent, serious sexually transmitted infection (e.g. gonorrhea, syphilis, chlamydia).
7. Currently using condoms for protection against a known sexually transmitted infection.
8. Taking any internally applied medication or oral medication to treat a genital condition.
9. Male partner has had difficulty achieving or maintaining an erection, or achieving ejaculation in the last month under typical circumstances/conditions.
10. Any self-reported genital condition (e.g. itching, burning, irritation, etc.) which, in the opinion of the investigator, could affect use of the study condoms or the ability to interpret study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We are recruiting heterosexual couples: 1 female and 1 male
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
User Preference to demonstrate feasibility of the prototoype | 2-3 weeks
  Couples comparing the comfort, lubrication, and experience with the HydroGlyde condom to a US leading silicone lubricated condom control. Couples will provide their feedback and experience in an online questionnaire and report which sample is most preferred.

CONTACTS AND LOCATIONS:
Locations (1):
- Essential Access Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
All information will only be shared by the sponsor (HydroGlyde Coatings, LLC) and clinical investigator (Essential Access Health).